CLINICAL TRIAL: NCT02533830
Title: Gum Chewing And Bowel Motility in Patients Undergoing Cesarean Section. Kasr el Ainy Experience.A Randomized Controlled Trial
Brief Title: Gum Chewing And Bowel Motility in Patients Undergoing Cesarean Section. Kasr el Ainy Experience
Acronym: RCT
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Kasr El Aini Hospital (Other)
Responsible Party: Principal Investigator, Mohamed El-Sharkawy, Lecturer of obstetrics and gynecology, Kasr El Aini Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: KasrELAini hospital
Record Dates: First submitted 2015-08-21; First posted 2015-08-27 (Estimated); Last update posted 2016-02-01 (Estimated); Status verified 2015-08

CONDITIONS: Gum Chewing; Bowel Function

STUDY DESIGN:
Who Masked: Care Provider
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- gum chewing group. (Active Comparator): Group A (81 Women) Who Received One Stick of Sugarless Gum (Samara for food & Chocolates Product Company)"S.A.E." , for 15 Minutes Every 2 hours After Surgery Tell Defecation
  Interventions: Biological: sugarless gum
- Placebo group (Placebo Comparator): Group B (81 Women) had Traditional Management (Oral Intake of Clear Fluid Allowed After Passage of Flatus and Regular Diet With The Passage of Bowel Movement.
  Interventions: Other: traditional management

INTERVENTIONS:
Biological: sugarless gum — One Stick of Sugarless Gum (Samara for food & Chocolates Product Company)"S.A.E." , for 15 Minutes Every 2 hours After Surgery Tell Defecation
  Other Names: Samara Gum
  Arms: gum chewing group.
Other: traditional management — Traditional Management (Oral Intake of Clear Fluid Allowed After Passage of Flatus and Regular Diet With The Passage of Bowel Movement.
  Arms: Placebo group

SUMMARY:
The aim of the present study was to evaluate the effect of chewing gum on the recovery of bowel function after cesarean section in women.

DETAILED DESCRIPTION:
This study Will Be conducted on 162 Patients Undergoing caesarean section in The Obstetrics & Gynecology Department "kasr el ainy teaching hospital".

Methods:

Women Were Randomized into Two Groups: Group A (81 Women) Who Received One Stick of Sugarless Gum (Samara for food & Chocolates Product Company)"S.A.E." , for 15 Minutes Every 2 hours After Surgery Tell Defecation , Group B (81 Women) had Traditional Management (Oral Intake of Clear Fluid Allowed After Passage of Flatus and Regular Diet With The Passage of Bowel Movement.

Each Women in Both Groups Was Examined Abdominal Using A Stethoscope Detect The Intestinal Movement Every 4 Hours And Asked to Report Immediately The Time of Either Passing Flatus or stool .

ELIGIBILITY:
Inclusion Criteria:

1. Age between 18 - 35 Years.
2. Spinal Anesthesia.
3. Pfannenstiel incision.

Exclusion Criteria:

1. History of Drug Consumption Especially Opioids.
2. Water and Electrolyte Disturbances.
3. Pancreatitis.
4. Peritonitis.
5. History of Abdominal Surgery except Cesarean Section.
6. No Willingness to Cooperative.
7. Intra and Sever Post-Operative Complications.
8. Inability to Chew Gum with Drawl.
9. Diabetes.
10. Pre-eclampsia
11. Prolonged Rupture of Membranes.
12. Hypothyroidism.
13. Muscular and Neurological Disorders.

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 162 (Estimated)
Dates: Start 2015-08; Primary Completion 2016-07 (Estimated); Study Completion 2016-07 (Estimated)

PRIMARY OUTCOMES:
the first audible bowel sound in hours | 4 months
  The First Bowel Sounds (Hours) The First Passage of Flatus (Hours) The First Defection (Hours) The First Bowel Sounds (Hours) The First Passage of Flatus (Hours) The First Defection (Hours) the first auscultation of regular bowel sounds in hours

SECONDARY OUTCOMES:
patient satisfaction | 4 months
  Change From Baseline in Pain on the 11 point Short Pain Scale (SPS-11)

CONTACTS AND LOCATIONS:
Overall Officials: Kasr El Ainy, Study Chair — kasr el ainy street,cairo,egypt
Locations (2):
- Egypt (2):
  - Mohamed Abdel Aziz El Sharkawy, Cairo
  - Mohqmed El Sharkawy, Cairo